CLINICAL TRIAL: NCT04474184
Title: Development of a Novel Early Detection Test to Reduce Racial Disparities in Endometrial Cancer (EC) Mortality
Brief Title: Development of a New Early Detection Test to Reduce Racial Disparities in Endometrial Cancer (EC) Death Rates
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 19-001140; NCI-2020-04756 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Focus Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aim 1 (focus group) (Experimental): Participants attend a focus group over 2 hours about endometrial cancer including knowledge of abnormal uterine bleeding, post-menopausal bleeding, risk factors, sources of medical information, barriers to seeking gynecologic care, and acceptance of tampon self-collection for endometrial cancer detection.
  Interventions: Behavioral: Focus Group; Other: Survey Administration
- Aim 2 (vaginal kit) (Experimental): Participants receive a tampon kit for collection of vaginal samples.
  Interventions: Procedure: Biospecimen Collection; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Receive vaginal kit for biospecimen collection
  Arms: Aim 2 (vaginal kit)
Behavioral: Focus Group — Attend focus group
  Arms: Aim 1 (focus group)
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase I trial investigates the development of a new early detection test to reduce racial disparities in endometrial cancer death rates. DNA samples collected from a tampon may be able to be used to detect endometrial cancer. Studying information from focus groups and vaginal samples of African American and white women may help researchers develop a less invasive and painful test to detect endometrial cancer. The purpose of this trial is to perform a demonstration project of tampon self-collection, assess percentage of samples returned; total and endometrial derived DNA quantity and quality, preliminarily test previously validated DNA methylation markers that may discriminate endometrial cancer from normal endometrium in tampon specimens.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To conduct focus groups to elicit perceptions and knowledge among African American women (AAW) and white women (WW) concerning abnormal uterine bleeding (AUB)/post-menopausal bleeding (PMB), endometrial cancer (EC) risk factors, barriers to seeking medical evaluation, sources of medical information and acceptance and feasibility of tampon self-collection for laboratory testing.

II. To perform a demonstration project of tampon self-collection from 25 AAW and 25 WW with AUB/PMB in Jacksonville.

OUTLINE:

AIM 1: Participants attend a focus group over 2 hours about endometrial cancer including knowledge of abnormal uterine bleeding, post-menopausal bleeding, risk factors, sources of medical information, barriers to seeking gynecologic care, and acceptance of tampon self-collection for endometrial cancer detection.

AIM 2: Participants receive a tampon kit for collection of vaginal samples.

After completion of study enrollment, participants may be followed up annually for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* AIM 1: Self-identified white women (WW) or African American women (AAW) (will record Hispanic ethnicity)
* AIM 2: Self-reported history of abnormal uterine bleeding (AUB) or post-menopausal bleeding (PMB)

Exclusion Criteria:

* AIM 1: Women who do not identify as WW or AAW
* AIM 1: Women who are unable to speak and read English
* AIM 2: Prior hysterectomy
* AIM 2: Prior pelvic radiation or are unwilling to comply with instructions
* AIM 2: Pregnant women

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Differences in views on endometrial cancer (EC) risk between African American and white women and whether the former would be willing to participate in tampon testing (Aim 1) | Up to 12 months
  Survey data will be reported as frequencies and proportions to describe the sample. Survey data will also be used to aid in interpretation of the qualitative data as appropriate.
Total deoxyribonucleic acid (DNA) (Aim 2) | Up to 12 months
Endometrial DNA (Aim 2) | Up to 12 months
Detection of EC-specific methylation markers (Aim 2) | Up to 12 months
  Will test samples for top EC-specific DNA methylation markers using methylation-specific polymerase chain reaction and provide descriptive statistics for all measurements (mean, median, standard deviation). Will assess the percentage of samples that yield > 500 ng amplifiable DNA, which suffices for methylation assays.

CONTACTS AND LOCATIONS:
Overall Officials: Mark E Sherman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States